CLINICAL TRIAL: NCT07195305
Title: Radiofrequency Endometrial Ablation or Uterine Artery Embolization for Women With Adenomyosis-related Abnormal Uterine Bleeding Eligible for Hysterectomy: a Non-inferiority Randomized Clinical Trial Comparing Each Intervention to Hysterectomy
Brief Title: Radiofrequency Endometrial Ablation or Uterine Artery Embolization for Treatment of Adenomyosis-related Abnormal Uterine Bleeding
Acronym: ADENOTREAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: French Ministry of Social Affairs and Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2024/47
Record Dates: First submitted 2025-08-18; First posted 2025-09-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Abnormal Uterine Bleeding Due to Adenomyosis (Disorder)
Keywords: Radiofrequency endometrial ablation; Uterine artery embolization; Hysterectomy; Adenomyosis; Abnormal uterine bleeding
MeSH Terms: conditions — Adenomyosis; Metrorrhagia | interventions — Uterine Artery Embolization; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiofrequency endometrial ablation (Experimental): Radiofrequency endometrial ablation performed using NovaSure®
  Interventions: Procedure: Radiofrequency endometrial ablation
- Uterine artery embolization (Experimental): Uterine artery embolization carried out under the guidance of digital subtraction angiography
  Interventions: Procedure: Uterine artery embolization
- Hysterectomy (Active Comparator): Hysterectomy
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Radiofrequency endometrial ablation — Radiofrequency endometrial ablation
  Arms: Radiofrequency endometrial ablation
Procedure: Uterine artery embolization — Uterine artery embolization
  Arms: Uterine artery embolization
Procedure: Hysterectomy — Hysterectomy
  Arms: Hysterectomy

SUMMARY:
The present study aims to compare the efficacy (menstrual blood loss, pain, quality of life) and the safety (complications, recovery) of each conservative intervention (RFA, UAE) versus hysterectomy for the treatment of adenomyosis-related abnormal uterine bleeding, up to 2 years

DETAILED DESCRIPTION:
Adenomyosis is defined by the presence of ectopic non-atypical endometrial glands and stroma within the smooth muscle fibers of the myometrium causing reactive hypertrophy of the uterus. The prevalence of adenomyosis is approximately 20% before 40 years, and probably higher in the following decade. One-third of women with adenomyosis are symptomatic. Symptoms include abnormal uterine bleeding (AUB) (40-50%), pelvic pain (dysmenorrhea 15-30%, dyspareunia) and are related to the uniformly enlarged and globular uterus (distension, swelling). Adenomyosis can be diagnosed by transvaginal ultrasonography and/or magnetic resonance imaging (MRI). Symptoms associated with adenomyosis can be treated by hormonal or non-hormonal medications. When medical treatment fails, a hysterectomy is proposed to women who do not consider childbearing. For women who wish to preserve their uterus, two alternatives are possible.

Radiofrequency ablation (RFA) is intended to ablate the endometrial lining of the uterus on pre-menopausal women with AUB due to benign causes for whom childbearing is complete. This outpatient procedure is well tolerated, with 10% of post-operative adverse events within one year, mainly not serious like pelvic pain/cramping and vaginal discharge/infection.

Uterine artery embolization (UAE) is as a minimally invasive treatment for symptomatic uterine fibroids since 1995. This procedure is also well tolerated, with efficacy and satisfaction rates of 85% at 2 years, performed usually as a day case or with a short hospital stay of 12-24h to manage immediate post-operative pain.

Therefore the extension of the indications of both techniques in AUB associated with adenomyosis should be questioned.

The present study aims to compare the efficacy (menstrual blood loss, pain, quality of life) and the safety (complications, recovery) of each conservative intervention (RFA, UAE) versus hysterectomy for the treatment of adenomyosis-related abnormal uterine bleeding, up to 2 years

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 30 to 50 years
* Women who had at least 3 prior months failed medical therapy, or a contraindication to medical therapy, or refused medical therapy for adenomyosis-related AUB
* Symptomatic pure internal adenomyosis or dominant adenomyosis (with less than 5 concurrent uterine fibroids type 3-7 < 5 cm) confirmed by MRI (< 6 months) according to ESHRE criteria
* AUB defined as a PBAC score >100 at baseline
* Uterine ultrasound measurement of 6.0-12.0 cm (external os to internal fundus)
* Women with an indication for hysterectomy for adenomyosis-related AUB and accepting hysterectomy
* Highly effective contraception for women of childbearing potential, maintained until the onset of menopause
* Affiliated or beneficiary of health insurance
* Signed informed consent

Exclusion Criteria:

* Uterine cavity abnormality or obstruction confirmed via imaging modalities or hysteroscopy
* Deep infiltrating posterior subperitoneal endometriosis involving contiguous digestive tract structures
* Uterine malignancy within the last five years
* Secreting ovarian tumor
* Atypical endometrial hyperplasia
* Unaddressed high grade cervical intra-epithelial lesions
* Active sexually transmitted disease or pelvic inflammatory disease
* Documented or suspected coagulopathies or long-term blood-thinner medications
* Prior transmural myomectomy or prior endometrial ablation
* Plasma FSH level > 40 IU/mL
* Any contraindication to angiography (including iodine allergy and creatinine clearance < 60mL/min)
* Any contraindication to MRI (claustrophobia, pace maker, etc.)
* Any contraindication to the use of Embosphere®, Embozene® or NovaSure® according to the instruction for use
* Women who are pregnant, breastfeeding, or who are planning to become pregnant
* Any condition or any situation that would prohibit women from coming to the investigational center for the 6 months follow-up
* Women unable to understand the nature, risks, significance and implications of the clinical investigation
* Women under legal protection

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
proportion of 2-year clinical success of the intervention | Year 2
  proportion of 2-year clinical success of the intervention, defined as a significant reduction in menstrual blood loss (Pictorial Blood Assessment Chart-PBAC, score <100). Women undergoing RFA or UAE and requiring subsequent hysterectomy for persistent AUB before 2 years will be considered as clinical failure.

SECONDARY OUTCOMES:
Proportion clinical success of the intervention | Month 1, Month 5, Year 1
  Proportion clinical success of the intervention, defined as a significant reduction in menstrual blood loss (PBAC score <100)
Proportion in self-reported amenorrhea | Month 1, Month 5, Year 1, Year 2
  Proportion in self-reported amenorrhea (PBAC score = 0),
Mean changes in severity of dysmenorrhea between UAE and RFA | Year 2
  Mean changes in severity of dysmenorrhea between Uterine Artery Embolisation-UAE and Radiofrequency endometrial ablation-RFA) (visual analogue scale rating from 0 to 10),
Mean changes in pelvic pain | Year 2
  Mean changes in pelvic pain (visual analogue scale rating from 0-no pain to 10-extreme pain);
Mean changes in deep dyspareunia | Year 2
  Mean changes in deep dyspareunia (visual analogue scale rating from 0-no pain to 10-extreme pain);
Mean changes in pelvic distension | Year 2
  Mean changes in pelvic distension (visual analogue scale rating from 0-no pain to 10-extreme pain);
Mean duration of hospital stay | Hospital discharge
  Mean duration of hospital stay (in days);
Mean time to return to normal life | Month 1
  Mean time to return to normal life (in days);
Mean change in quality of life | Year 2
  Mean change in quality of life assessed using UFS-QoL questionnaire (Uterine Fibroid Symptom Health-Related Quality of Life Questionnaire, from 29 poins (best health-related quality of life to 145 (worse health-related quality of life)
Mean change in endometriosis quality of life | Year 2
  Mean change in endometriosis quality of life assessed using EHP-5 questionnaire (Short form endometriosis health profile, from 0 (best possible state of health) to 100 (worst possible state of health)
Mean change in sexual life quality | Year 2
  Mean change in sexual life quality using FSFI questionnaire (Female Sexual Function Index from 2 (worse sexual life quality to 36 (best sexual life quality; 26.55 indicating the lower score reflecting the existence of sexual disorders
Mean satisfaction with the intervention | Year 2
  Mean satisfaction with the intervention (7-point Likert scale) from hospital discharge to 2 years;
Proportion of women with correction of iron-deficiency anemia | Year 2
  Proportion of women with correction of iron-deficiency anemia, if diagnosed at baseline
Rate and severity of intra-operative complications | Hospital discharge
  Rate and severity of intra-operative complications (according to Clavien Dindo classification)
Severity of intra-operative complications | Hospital discharge
  Severity of intra-operative complications (according to Clavien Dindo classification)
Analgesic and/or non-steroidal anti-inflammatory drug intake | Week 1
  Analgesic and/or non-steroidal anti-inflammatory drug intake (type, daily dose, duration)
Rate of post-operative adverse events | Year 2
  Rate of post-operative adverse events
Severity of post-operative adverse events | Year 2
  Severity of post-operative adverse events
Mean change in junctional zone thickness | Month 6
  Mean change in MRI junctional zone thickness accordingly to European Society of Human Reproduction and Embryology-ESHRE- criteria bewteen Uterine Artery Embolisation-UAE and Radiofrequency endometrial ablation-RFA
Mean change in percentage of necrosis | Month 6
  Mean change in MRI percentage of necrosis accordingly to European Society of Human Reproduction and Embryology-ESHRE- criteria bewteen Uterine Artery Embolisation-UAE and Radiofrequency endometrial ablation-RFA
Mean change in uterine vascularization | Month 6
  Mean change in MRI uterine vascularization accordingly to European Society of Human Reproduction and Embryology-ESHRE- criteria bewteen Uterine Artery Embolisation-UAE and Radiofrequency endometrial ablation-RFA
Mean change of hormonal parameters | Year 2
  Mean change of hormonal parameters (FH, estradiol), if post-operative amenorrhea occurred after Uterine Artery Embolisation-UAE and Radiofrequency endometrial ablation-RFA

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No